CLINICAL TRIAL: NCT00728611
Title: PRP as a Treatment for Knee Osteoarthritis - Randomized-double-blind-placebo Control Trail.
Brief Title: Preparation Rich in Growth Factors (PRGF) Treatment for Osteoarthritis of the Knee
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Meir Medical Center (Other)
Responsible Party: Omer Mei Dan, Meir Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1000
Record Dates: First submitted 2008-08-03; First posted 2008-08-06 (Estimated); Last update posted 2011-07-12 (Estimated); Status verified 2011-07

CONDITIONS: Osteoarthritis of the Knee
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Intercellular Signaling Peptides and Proteins; Hyaluronic Acid; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Experimental)
  Interventions: Biological: PRGF
- 2 (Active Comparator)
  Interventions: Drug: hyaluronic acid
- 3 (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Biological: PRGF — intra auricular injection 6mg
  Other Names: platelet-derived preparation rich in growth factors
  Arms: 1
Drug: hyaluronic acid — 20 mg / 2 ml
  Other Names: Arthrease
  Arms: 2
Drug: placebo — physiological water 3cc + lidocain 3cc
  Other Names: seline 0.9% nacl
  Arms: 3

SUMMARY:
to evaluate the influence of PRGF treatment on patient suffering from OA knee

DETAILED DESCRIPTION:
Autologous platelet-secreted growth factors (GFs) may have therapeutic effects in osteoarthritis (OA) capsular joints via multiple mechanisms. Our aim is to examine the effect of a platelet-derived preparation rich in growth factors (PRGFs) in OA knee

ELIGIBILITY:
Inclusion Criteria:

* age 40-75 years old
* diagnosed Oa of the knee more then 1 year
* no knee deformation

Exclusion Criteria:

* mental of physical disabilities
* pregnancy
* deformities of the knee

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2008-01; Primary Completion 2009-02 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Improvment of symptomes | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Meir Medical Center, Kfar Saba, Israel